CLINICAL TRIAL: NCT06343493
Title: Effect of Hot Saline Irrigation on the Operative Field During Endoscopic Sinus Surgery: A Randomized Controlled Trial
Brief Title: Effect of Hot Saline Irrigation on the Operative Field During Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, JAWAIRIA ALTAF, Postgraduate trainee ENT, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JALTAF
Record Dates: First submitted 2024-03-17; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Rhinosinusitis
Keywords: Endoscopic sinus surgery; Operative field; Saline
MeSH Terms: conditions — Rhinosinusitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Interventional Group) (Experimental): Hot saline with a temperature of 50°C used for irrigation during endoscopic sinus surgery. Frequency of the drug is according to the operative field and surgeon's need.
  Interventions: Drug: Normal saline heated up to 50 °C
- Group B (Control Group) (No Intervention): Saline at room temperature used for irrigation during endoscopic sinus surgery. Frequency according to the operative field and surgeon's need.

INTERVENTIONS:
Drug: Normal saline heated up to 50 °C — Saline heated up to 50 °C used for irrigation
  Other Names: NaCl 0.9%
  Arms: Group A (Interventional Group)

SUMMARY:
Control of bleeding is very important during endoscopic sinus surgery. Saline heated up to 50°C causes dilatation of vessels and edema without nasal mucosa necrosis. It also promotes the clotting cascade so helps in having a bloodless procedure.

This randomized controlled trial was conducted on 60 patients divided into two groups (30 each). Group A was the interventional group in which patients were irrigated with saline of 50°C during surgery. Group B was the control group where room temperature saline was used. Operative field was assessed using the Boezaart score, duration of surgery and bleeding in ml.

KEY WORDS:

* Chronic rhinosinusitis (CRS)
* Endoscopic sinus surgery
* Boezaart score

DETAILED DESCRIPTION:
INTRODUCTION: Chronic rhinosinsusitis is an inflammatory disease of the sinonasal mucosa lasting for more than 12 weeks. Endoscopic sinus surgery is the surgical procedure used to treat recalcitrant chronic rhinosinusitis. It not only helps in the drainage of sinuses and removal of pathology but also prevents the disturbance of anatomy and formation of facial scars. Control of bleeding during the procedure is a test for surgeons as well as anesthetists. Capillaries are the commonest vessels to bleed during the surgery so that's why mean arterial pressure is an important determinant of the severity of bleeding. A good control of bleeding gives a good visualization of the anatomy during the procedure.

There are different ways to reduce bleeding but all carry side effects too. Topical vasoconstrictors may also be absorbed systemically so must be used carefully in children and patients with cardiac ischemia. Moreover, there's no accurate way to measure absorption of a vasoconstrictor so it's difficult to recommend a safe dose for a particular patient. Cautery which is used to seal blood vessels is also associated with pain as well as mucosal damage. Anesthesia induced hypotension is also not appropriate for all patients as it results in decreased oxygen supply to various vitals organs of the body.

Normal saline heated up to 50°C causes dilatation of vessels and nasal edema without causing nasal mucosa necrosis. This edema compresses blood vessels and helps in controlling bleeding. It also promotes the clotting cascade. In addition, it provides better visualization of the surgical field by reduction of fog formation. A study conducted by Shehata A et al. showed a significant improvement in the operative field when normal saline at 50° C was used during endoscopic sinus surgery. Not only the operative filed was improved, also the duration of surgery was significantly reduced. According to the results of this study, saline heated up to 50°C used for the irrigation of endoscopic sinus surgery produced a result comparable to usage of tranexamic acid with a significant p value. Another study by Ranford D et al. concluded that irrigation with heated saline during endoscopic sinus surgery reduced bleeding by 20 percent.

This study aims to assess the effect of heated normal saline up to 50°C upon the operative field during endoscopic sinus surgery. The use of hot saline for irrigation during endoscopic sinus surgery can prove to be a cost effective method to have a bloodless field during surgery.

METHODS AND MATERIALS:

This randomized controlled trial was conducted after approval from the ethical board in the setting of department of ENT and head & neck surgery, Benazir Bhutto Hospital, Rawalpindi over a period of ten months from June 2023 to Dec 2023. The sampling technique was simple random sampling. The patients were divided into two groups (treatment group and control group) via randomization using the lottery method. Sample size came out to be 60, with 30 patients in each group. Proper written consents taken from the patients and the surgery was done in the ENT operation theatre by a surgeon with an experience of more than 5 years.

Patient with bilateral chronic rhinosinusitis and pansinusitis on plain CT scan nose and paranasal sinuses were included in the study. Patients with unilateral disease, uncontrolled hypertension, diabetes or other significant comorbidities were excluded. Moreover, patients with the suspicion of malignancy, CSF leak and bleeding diathesis affecting the results were also not included in the study. Group A was the interventional group in which normal saline heated up to 50°C was irrigated during surgery. Normal saline was heated in a boiler and a temperature of 50°C was continuously maintained and monitored. Mean arterial pressure appropriate for endoscopic sinus surgery was controlled by the anesthetist using different drugs for hypotensive anesthesia and it was recorded after every 15 minutes. Intra-operative blood loss was measured from the glass suction tank after subtraction of the irrigated normal saline.

The patient, operating surgeon and primary investigator were blinded during the study to prevent bias. To assess the operative field, subjective grading was done by the surgeon using the Boezaart score. Wait and watch approach was followed to assess bleeding control. Total duration of surgery was also recorded. At the end of the surgery, bilateral anterior nasal packing was done.

ANALYSIS PLAN:

The data was analysed by SPSS version 26. Quantitative data was expressed as mean and standard deviation. Qualitative data was represented as frequencies and percentages. Independent sample T tests was used for the quantitative data analysis. Moreover different correlations were done via Spearman and Kendall test. A P value of <0.05 was considered as significant and a P value of <0.001 showed a high significance.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic rhinosinusitis requiring surgery

Exclusion Criteria:

* Unilateral disease
* Suspicion of malignancy
* CSF leak
* Bleeding diathesis
* Significant comorbidities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Boezaart Score | Per operative
  Operative field is assessed based on the Boezaart score which is a subjective score graded from 0 to 5 where 0 shows no bleeding and is the minimum score. 5 is the maximum score which shows severe bleeding. So the outcome worsens as the grade becomes higher from 0 to 5. 5 shows the worst outcome.

SECONDARY OUTCOMES:
Bleeding in ml | Per operative
  Operative field assessed on the basis of blood loss in ml measured from the suction tanks after subtracting the irrigated saline volume
Duration of Surgery | From the start of surgery to the end (per operative)
  If the operative field is good, duration of surgery is decreased and vice versa

CONTACTS AND LOCATIONS:
Overall Officials: Jawairia Altaf PGR, Principal Investigator — Rawalpindi Medical College
Locations (1):
- Benazir Bhutto Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ranford D, Fu B, Surda P, Rudd J. Hot saline irrigation for haemostasis in functional endoscopic sinus surgery: a systematic review and meta-analysis. J Laryngol Otol. 2022 Aug;136(8):676-682. doi: 10.1017/S0022215121003698. Epub 2021 Nov 25. PMID 34819186
- [Result] Dalziel K, Stein K, Round A, Garside R, Royle P. Endoscopic sinus surgery for the excision of nasal polyps: A systematic review of safety and effectiveness. Am J Rhinol. 2006 Sep-Oct;20(5):506-19. doi: 10.2500/ajr.2006.20.2923. PMID 17063747
- [Result] Senior BA, Kennedy DW, Tanabodee J, Kroger H, Hassab M, Lanza D. Long-term results of functional endoscopic sinus surgery. Laryngoscope. 1998 Feb;108(2):151-7. doi: 10.1097/00005537-199802000-00001. PMID 9473061

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT06343493/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT06343493/ICF_001.pdf